CLINICAL TRIAL: NCT00357162
Title: Phase II Study of the Histone Deacetylase Inhibitor PXD101 for the Treatment of Myelodysplastic Syndrome
Brief Title: Belinostat in Treating Patients With Myelodysplastic Syndromes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00143; NCI-2009-00143 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MAYO-MC0581; NCI-7258; CDR0000489197; MC0581 (Other: Mayo Clinic); 7258 (Other: CTEP); P30CA015083 (NIH); N01CM62205 (NIH); NCT01647009 (obsolete NCT alias); NCT01664429 (obsolete NCT alias)
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Results first posted 2013-03-20 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2011-12

CONDITIONS: de Novo Myelodysplastic Syndromes; Previously Treated Myelodysplastic Syndromes; Secondary Myelodysplastic Syndromes
MeSH Terms: interventions — belinostat

ARMS (1):
- Treatment (enzyme inhibitor therapy) (Experimental): Patients receive belinostat IV over 30 minutes on days 1-5. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: belinostat

INTERVENTIONS:
Drug: belinostat — Given IV
  Other Names: PXD101

SUMMARY:
This phase II trial is studying how well belinostat works in treating patients with myelodysplastic syndromes. Belinostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Establish the efficacy and safety of PXD101 (belinostat) in patients with myelodysplastic syndromes that progressed after or is ineligible for azacitidine treatment.

II. Assess the biological activity of PXD101 in these patients via assays of histone acetylation, gene expression profiling, and DNA methylation.

OUTLINE: This is a multicenter study.

Patients receive belinostat intravenously (IV) over 30 minutes on days 1-5. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients achieving complete response, partial response, or hematologic improvement after 4 courses receive 4 additional courses of therapy. After completion of study treatment, patients are followed every 3-6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed myelodysplastic syndromes (MDS)

  * De novo or secondary MDS
* Patients with < 5 % bone marrow blasts must meet ≥ 1 of the following criteria:

  * Symptomatic anemia with either hemoglobin < 10.0 g/dL or required RBC transfusions within the past 3 months
  * Thrombocytopenia with ≥ 2 platelet counts < 50,000/mm³ or significant hemorrhage requiring platelet transfusions
  * Neutropenia with ≥ 2 absolute neutrophil counts < 1,000/mm³
* No acute myeloid leukemia (≥ 20% bone marrow blasts)
* ECOG performance status 0-2
* Life expectancy > 12 weeks
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST ≤ 2 times ULN
* Creatinine ≤ 2.0 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to PXD101
* No HIV positivity
* QTc interval ≤ 500 msec
* No long QT syndrome
* No significant cardiovascular disease, including any of the following:

  * Unstable angina pectoris
  * Uncontrolled hypertension
  * Congestive heart failure related to primary cardiac disease
  * Condition requiring anti-arrhythmic therapy
  * Ischemic or severe valvular heart disease
  * Myocardial infarction within the past 6 months
* No other uncontrolled serious medical condition (e.g., cardiac arrhythmias or diabetes)
* Recovered from prior therapy
* No more than 2 prior therapies for MDS

  * Prior hematopoietic growth factors, androgens, and other supportive care agents allowed and are not considered in the prior therapy total
* No prior allogeneic stem cell transplantation
* More than 4 weeks since prior radiotherapy or chemotherapy (6 weeks for nitrosoureas or mitomycin C)
* No prior histone deacetylase (HDAC) inhibitors for treatment of MDS
* More than 2 weeks since prior valproic acid or other HDAC inhibitors
* No other concurrent investigational agents
* No concurrent medication that may cause torsades depointes, including any of the following:

  * Disopyramide
  * Dofetilide
  * Ibutilide
  * Procainamide
  * Quinidine
  * Sotalol
  * Bepridil
  * Methadone
  * Amiodarone hydrochloride
  * Arsenic trioxide
  * Cisapride
  * Calcium-channel blockers (e.g., lidoflazine)
  * Anti-infective agents (i.e., clarithromycin, erythromycin, halofantrine, pentamidine, or sparfloxacin)
  * Domperidone or droperidol
  * Antipsychotic agents (i.e., chlorpromazine, haloperidol, mesoridazine, thioridazine, or pimozide)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Cashen, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-one patients were accrued, and all were eligible and> evaluable.
Period: Overall Study
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 67 [48 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Confirmed Responses (Complete Response, Partial Response, or Hematologic Improvement) Noted on 2 Consecutive Evaluations at Least 4 Weeks Apart
Description: Complete Response (CR)
  A CR is defined as a participant with bone marrow showing less than 5% myeloblasts with no evidence of dysplasia and with adequate peripheral blood counts for at least 2 months (hemoglobin > 11 g/dl, neutrophils ≥ 1500/mm3, platelets ≥ 100,000/mm3) and with no blasts in the peripheral.
  Partial Response (PR)
  All the CR criteria except bone marrow blasts decreased by ≥ 50% over pretreatment, or a less advanced WHO classification than pretreatment.
  Hematologic Improvement (HI)
  A 2g/dl increase in hemoglobin for participants with <11g/dl hemoglobin at pretreatment, or an increase of >30,000/mm^3 platelets for participants with <100,000/mm^3 at pretreatment, or a 100% increase in neutrophil counts for participants with <1500/mm^3 at pretreatment
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 21
participants
  Confirmed Hematologic Improvement (HI) | 1
  Confirmed Partial Response (PR) | 0
  COnfirmed Complete Response (CR) | 0

2. Secondary Outcome: Time to Progression
Description: Estimated using the method of Kaplan-Meier.
Time Frame: Time from registration to the date of progression or last follow-up, assessed up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 21
months | 14.9 [5.8 to 30]

3. Secondary Outcome: Overall Survival
Description: Estimated using the method of Kaplan-Meier.
Time Frame: From date of registration to the date of last follow-up or death due to any cause, assessed up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 13
months | 17.9 [13.2 to 30]

4. Secondary Outcome: Duration of Response
Description: Estimated using the method of Kaplan-Meier.
Time Frame: From the date of documented response until the date of progression or last follow-up, assessed up to 3 years
Population: One participant had a confirmed Hematologica Improvement. For patient confidentiality, we are not reporting response data.
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 0

5. Secondary Outcome: Toxicity of Belinostat in Patients With Myelodysplastic Syndrome
Description: Graded using the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. Reporting events deemed at least possibly related to study treatment.
Time Frame: Prior to each course (every 21 days), and every 3 months for up to 3 years after completion of study treatment
Measure: Number; unit: participants
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 21
participants
  Grade 3 Hematologic Adverse Event | 13
  Grade 4 Hematologic Adverse Events | 11
  Grade 3 Non-Hemeatologic Adverse Events | 5
  Grade 4 Non-hematologic Adverse Events | 1

ADVERSE EVENTS:
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Serious Adverse Events (participants affected / at risk) | 10/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Enzyme Inhibitor Therapy) (N=21)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Disease progression (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 3 (3)
Neutrophil count decreased (Investigations) | 5 (6)
Platelet count decreased (Investigations) | 4 (7)
Syncope (Nervous system disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Enzyme Inhibitor Therapy) (N=21)
Hemoglobin decreased (Blood and lymphatic system disorders) | 20 (100)
Left ventricular failure (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 7 (15)
Diarrhea (Gastrointestinal disorders) | 6 (18)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 17 (34)
Vomiting (Gastrointestinal disorders) | 7 (10)
Edema limbs (General disorders) | 3 (5)
Fatigue (General disorders) | 19 (64)
Fever (General disorders) | 1 (1)
Injection site reaction (General disorders) | 2 (5)
Cytokine release syndrome (Immune system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 2 (3)
Infection (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 5 (17)
Alkaline phosphatase increased (Investigations) | 1 (3)
Aspartate aminotransferase increased (Investigations) | 4 (6)
Blood bilirubin increased (Investigations) | 2 (4)
Creatinine increased (Investigations) | 1 (1)
Electrocardiogram QTc interval prolonged (Investigations) | 2 (2)
Leukocyte count decreased (Investigations) | 19 (71)
Lymphocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 18 (62)
Platelet count decreased (Investigations) | 18 (73)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Blood glucose increased (Metabolism and nutrition disorders) | 4 (7)
Iron overload (Metabolism and nutrition disorders) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 1 (1)
Serum calcium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (3)
Serum magnesium decreased (Metabolism and nutrition disorders) | 1 (2)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum sodium increased (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Dizziness (Nervous system disorders) | 4 (6)
Dysgeusia (Nervous system disorders) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 5 (9)
Anxiety (Psychiatric disorders) | 1 (1)
Confusion (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (3)
Kidney pain (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (15)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (2)
Sweating (Skin and subcutaneous tissue disorders) | 1 (2)
Flushing (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less